CLINICAL TRIAL: NCT02930590
Title: Comparing the Effects of Three Different Support Surfaces on the Properties of Heel and Sacral Skin After Loading
Brief Title: Effects of Different Support Surfaces on the Properties Skin After Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jan Kottner, PD Dr., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: CRC-PU-A-23
Record Dates: First submitted 2016-09-26; First posted 2016-10-12 (Estimated); Results first posted 2018-10-23 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-05

CONDITIONS: Pressure Ulcers
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Pressure mattress (Experimental): Alternating Low Pressure mattress with low air loss function (IsoAir, stryker, USA)
  Interventions: Other: Alternating low pressure mattress with air loss function
- Reactive support surface (Experimental): Gel mattress (IsoGel, stryker, USA)
  Interventions: Other: Gel mattress
- Standard mattress (Active Comparator): basic foam
  Interventions: Other: Basic foam

INTERVENTIONS:
Other: Alternating low pressure mattress with air loss function — IsoAir, Stryker, USA
  Arms: Low Pressure mattress
Other: Gel mattress — IsoGel, Stryker, USA
  Arms: Reactive support surface
Other: Basic foam — Standard hospital mattress
  Arms: Standard mattress

SUMMARY:
Pressure ulcers are severe injuries and wounds causing a substantial burden on patients, caregivers, and on healthcare systems worldwide. There is common agreement, that effective pressure ulcer prevention is of crucial importance to maintain skin and tissue integrity in individuals at risk. Besides risk assessment and repositioning the use of special pressure ulcer preventive support surfaces are the key interventions in pressure ulcer prevention. Pressure ulcer preventive support surface modify the degree of skin and tissue deformation and/or skin temperature and moisture. Therefore, an association between the type and working mechanism of a pressure ulcer support surface and skin function after loading is highly likely. Furthermore, such a relationship may be used to characterize and/or to quantify the performance pressure ulcer support surfaces in terms of skin protection. The overall aim of this explorative study is to measure skin responses of the two most common pressure ulcer predilection sites (heel, sacral skin) after two hours loading on three different support surfaces and the sternal skin (control area).

ELIGIBILITY:
Inclusion Criteria:

* Healthy, female volunteers
* 60 to 80 years
* Body Mass Index between 18.5 and 29.9 kg/m2
* Non-Smoker of at least one year
* Absence of skin diseases or scars in the skin areas of interest
* Ability to move independently and to maintain supine and prone positions
* Able to give written informed consent
* No use of cosmetic products or topical applied drugs on the study areas at least 12 hours before measurement
* Skin phototype I to III according to Fitzpatrick classification
* Willing and able to fulfil the study requirements

Exclusion Criteria:

* Disability to maintain in supine or prone position
* Acute diseases
* Acute or chronic diseases with increased or decreased body temperature (≤ 35°C or ≥ 38,5°C, measured in the ear)
* History or establishment of Diabetes or pre-diabetes, cardiac or renal insufficiency, atopic dermatitis, psoriasis, chronic obstructive pulmonary disease (COPD)
* Acute or chronic wounds in the skin areas of interest
* Any skin affection which may interfere with the study assessment, e.g. tattoo, psoriasis or scar on the investigational sites
* Participation in another clinical study 4 weeks before inclusion visit
* Current participation in any other clinical study

Ages: 60 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kottner, PD Dr., Study Director — Charite University, Berlin, Germany
Locations (1):
- Charité-Universitätsmedizin Berlin, Berlin, Germany

REFERENCES:
- [Result] Tomova-Simitchieva T, Lichterfeld-Kottner A, Blume-Peytavi U, Kottner J. Comparing the effects of 3 different pressure ulcer prevention support surfaces on the structure and function of heel and sacral skin: An exploratory cross-over trial. Int Wound J. 2018 Jun;15(3):429-437. doi: 10.1111/iwj.12883. Epub 2017 Dec 26. PMID 29277963

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at the Clinical Research Center for Hair and Skin Science in Berlin, Germany from September 2016 to March 2017 and involved 15 healthy female volunteers.
Groups:
- Low Pressure, Reactive Support, Than Standard Mattress; Low Pressure, Standard Mattress, Than Reactive Support; Reactive Support, Low Pressure, Than Standard Mattress; Reactive Support, Standard Mattress, Than Low Pressure; Standard Mattress, Low Pressure, Than Reactive Support; Standard Mattress, Reactive Support, Than Low Pressure: Alternating Low Pressure Mattress with Low Air Loss Function (IsoAir, Stryker, USA) Reactive Support Surface: Gel mattress (IsoGel, Stryker, USA) Standard Mattress: Basic foam (Stryker, USA)
Period: First Intervention (2 Hours)
Arm/Group | Low Pressure, Reactive Support, Than Standard Mattress | Low Pressure, Standard Mattress, Than Reactive Support | Reactive Support, Low Pressure, Than Standard Mattress | Reactive Support, Standard Mattress, Than Low Pressure | Standard Mattress, Low Pressure, Than Reactive Support | Standard Mattress, Reactive Support, Than Low Pressure
Started (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Completed (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Hours)
Arm/Group | Low Pressure, Reactive Support, Than Standard Mattress | Low Pressure, Standard Mattress, Than Reactive Support | Reactive Support, Low Pressure, Than Standard Mattress | Reactive Support, Standard Mattress, Than Low Pressure | Standard Mattress, Low Pressure, Than Reactive Support | Standard Mattress, Reactive Support, Than Low Pressure
Started (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Completed (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Hours)
Arm/Group | Low Pressure, Reactive Support, Than Standard Mattress | Low Pressure, Standard Mattress, Than Reactive Support | Reactive Support, Low Pressure, Than Standard Mattress | Reactive Support, Standard Mattress, Than Low Pressure | Standard Mattress, Low Pressure, Than Reactive Support | Standard Mattress, Reactive Support, Than Low Pressure
Started (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Completed (Cross-over trial.In total 15 participants,each of them lied on every of the three types of mattress.) | 3 | 3 | 3 | 2 | 2 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross-over trial. In total 15 participants, each of them lied on every of the three types of mattress.
Groups:
- AlternatingLow Pressure Mattress,Reactive Mattress,Basic Foam: Cross-over trial. In total 15 participants, each of them lied on every of the three types of mattress.
Arm/Group | AlternatingLow Pressure Mattress,Reactive Mattress,Basic Foam
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 66 [63 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 15
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m2] | 24.5 [23.7 to 26.0]
Body temperature [Median (Inter-Quartile Range); unit: °C] | 36.3 [36.3 to 36.6]
Heart rate [Median (Inter-Quartile Range); unit: beats per minute] | 78 [66 to 80]
Systolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 125 [115 to 140]
Diastolic blood pressure [Median (Inter-Quartile Range); unit: mmHg] | 75 [70 to 85]
Skin phototype [Count of Participants; unit: Participants] — Assessment of the participants' skin phototype according Fitzpatrick classification with six categories. Participants with the skin phototype I (celtic type: fair ivory skin, red or blond hair, blue eyes and freckles; tans never, burns always), II (fair "caucasian": white skin, blond hair, blue or green eyes; tans a little, burns easily) and III (dark "caucasian": white skin, brown hair, gray or brown eyes; tans moderately, burns moderately) have been included in this study.
  Participants
    Skin phototype I | 3
    Skin phototype II | 9
    Skin phototype III | 3

OUTCOME MEASURES:

1. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Sacrum, at Baseline
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: at baseline
Population: Cross-over trial with 15 female participants between 60 and 80 years, each of them lied on every of the three types of mattress.
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Groups:
- Alternating Low Pressure Mattress: Alternating Low Pressure mattress with low air loss function (IsoAir, Stryker, USA)
  Alternating low pressure mattress with air loss function: IsoAir, Stryker, USA
- Standard Mattress: Basic foam (Stryker, USA)
  Basic foam: Standard mattress, Stryker, USA
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 7.8 [6.7 to 8.8] | 7.7 [6.7 to 8.2] | 7.1 [6.8 to 8.8]

2. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Sacrum, After Two Hours Loading
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 12.4 [11.5 to 15.2] | 10.4 [8.5 to 12.2] | 14.5 [9.3 to 20.5]

3. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Sacrum, 20 Min After Off-loading
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 8.0 [7.0 to 8.6] | 7.6 [6.4 to 8.6] | 8.0 [6.8 to 9.0]

4. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Heel, at Baseline
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 8.1 [7.6 to 10.9] | 9.4 [8.2 to 11.6] | 8.6 [7.4 to 12.1]

5. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Heel, After Two Hours Loading
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 19.5 [16.6 to 25.3] | 19.2 [16.3 to 23.3] | 28.4 [15.9 to 32.3]

6. Primary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Heel, 20 Min After Off-loading
Description: TEWL was measured using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 9.6 [9.0 to 11.2] | 10.4 [8.9 to 13.3] | 11.1 [9.9 to 14.8]

7. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Sacrum, at Baseline
Description: Skin thermometer based on the infrared technique (Courage & Khazaka electronic GmbH, Cologne, Germany) was used to measure the skin surface temperature in °C.
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 28.8 [28.2 to 29.2] | 28.9 [28.3 to 29.2] | 29.1 [28.1 to 29.8]

8. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Sacrum, After Two Hours
Description: as for outcome 7
Time Frame: after two hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 31.4 [31.3 to 32.0] | 30.7 [30.5 to 31.3] | 32.0 [31.3 to 32.2]

9. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Sacrum, 20 Minutes After Off-loading
Description: as for outcome 7
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 30.3 [29.8 to 30.6] | 29.4 [29.2 to 30.1] | 30.3 [29.8 to 31.1]

10. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Heel, at Baseline
Description: as for outcome 7
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 24.4 [24.1 to 25.2] | 25.2 [24.3 to 25.4] | 24.3 [23.3 to 25.4]

11. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Heel, After Two Hours Loading
Description: as for outcome 7
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 26.5 [25.4 to 26.9] | 25.5 [24.7 to 26.2] | 26.6 [25.5 to 27.3]

12. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Heel, 20 Minutes After Off-loading
Description: as for outcome 7
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 25.4 [24.9 to 26.0] | 25.2 [23.8 to 25.4] | 25.9 [24.9 to 26.6]

13. Secondary Outcome: Erythema Index in Arbitrary Units at the Sacrum, at Baseline
Description: Erythema was measured with the Mexameter® MX 18 device by using specific wavelengths (the intensity of the reflected red (λ = 660 nm) and green (λ = 568 nm) lights) to measure the absorption capacity of the skin (specifically the content of hemoglobin in the skin). Lower values represent less redness.
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 187.5 [164.4 to 224.3] | 176.5 [142.7 to 211.1] | 167.2 [150.5 to 193.7]

14. Secondary Outcome: Erythema Index in Arbitrary Units at the Sacrum, After Two Hours Loading
Description: as for outcome 13
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 220.2 [185.0 to 251.4] | 206.0 [153.2 to 238.5] | 235.9 [191.3 to 275.2]

15. Secondary Outcome: Erythema Index in Arbitrary Units at the Sacrum, 20 Min After Off-loading
Description: as for outcome 13
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 201.3 [177.8 to 233.5] | 194.0 [147.0 to 218.5] | 221.0 [191.4 to 239.9]

16. Secondary Outcome: Erythema Index in Arbitrary Units at the Heels, at Baseline
Description: as for outcome 13
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 194.5 [132.2 to 225.4] | 177.9 [143.2 to 250.9] | 186.2 [116.7 to 234.7]

17. Secondary Outcome: Erythema Index in Arbitrary Units at the Heels, After Two Hours Loading
Description: as for outcome 13
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Groups:
- Standard Mattress: Basic foam (IsoGel, Stryker, USA)
  Basic foam: Standard mattress, Stryker, USA
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 247.1 [146.9 to 279.2] | 225.7 [160.0 to 272.5] | 225.2 [183.5 to 290.5]

18. Secondary Outcome: Erythema Index in Arbitrary Units at the Heels, 20 Min After Off-loading
Description: as for outcome 13
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 231.9 [145.9 to 246.0] | 188.5 [142.8 to 236.0] | 226.7 [143.7 to 246.9]

19. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Sacrum, at Baseline
Description: Corneometer® CM 825 (Courage & Khazaka electronic GmbH, Cologne, Germany) was used to measure SCH in arbitrary units (AU) (range 0-120 AU). Lower values represent reduced skin hydration in the upper skin layer.
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 27.2 [19.7 to 34.7] | 23.8 [19.5 to 35.8] | 27.5 [25.1 to 36.2]

20. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Sacrum, After Two Hours Loading
Description: as for outcome 19
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 34.6 [25.3 to 40.4] | 29.8 [22.0 to 40.0] | 31.6 [26.1 to 42.5]

21. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Sacrum, 20 Min Off-loading
Description: Corneometer® CM 825 (Courage & Khazaka electronic GmbH, Cologne, Germany) was used to measure SCH in arbitrary units (AU) (range 0-120 AU).Lower values represent reduced skin hydration in the upper skin layer.
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 29.3 [25.6 to 35.9] | 27.4 [22.7 to 36.4] | 30.1 [23.9 to 39.6]

22. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Heels, at Baseline
Description: as for outcome 21
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 13.3 [8.3 to 19.2] | 13.6 [9.3 to 21.1] | 12.9 [8.7 to 17.8]

23. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Heels, After Two Hours Loading
Description: as for outcome 19
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 18.0 [13.9 to 23.4] | 17.9 [12.5 to 23.4] | 20.2 [14.5 to 24.6]

24. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Heels, 20min Off-loading
Description: as for outcome 19
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 14.4 [10.7 to 22.1] | 12.9 [8.3 to 19.2] | 15.3 [10.8 to 17.8]

25. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Sacrum, at Baseline
Description: Skin roughness was measured using the Visioscan VC98 (Courage+Khazaka, Cologne, Germany) device. It consists of a UV light camera and measures the skin surface profiles. Rz is the arithmetic average of different segment roughness values calculated with visioscan software. The median was calculated from the Rz values from the 15 participants for each Intervention Group.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 39.5 [33.5 to 41.0] | 35.5 [33.3 to 44.6] | 34.0 [32.0 to 41.5]

26. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Sacrum, After Two Hours Loading
Description: as for outcome 25
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 39.0 [36.0 to 43.5] | 40.0 [37.0 to 43.5] | 39.5 [34.0 to 44.0]

27. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Sacrum, 20 Min After Off-loading
Description: as for outcome 25
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 43.0 [38.5 to 50.5] | 40.5 [36.0 to 49.0] | 42.5 [37.0 to 46.0]

28. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Sacrum, at Baseline
Description: Skin roughness was measured using the Visioscan VC98 (Courage+Khazaka, Cologne, Germany). It consists of a UV light camera and measures the skin surface profiles. Ra is the arithmetical mean roughness calculated with visioscan software. The median was calculated from the Ra values from the 15 participants for each Intervention Group.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 9.0 [8.0 to 10.0] | 8.3 [6.9 to 10.1] | 8.0 [7.5 to 10.0]

29. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Sacrum, After Two Hours Loading
Description: as for outcome 28
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 9.0 [8.0 to 11.5] | 9.0 [8.5 to 10.0] | 8.5 [7.5 to 10.0]

30. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Sacrum, 20 Min Off-loading
Description: as for outcome 28
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 10.0 [8.5 to 12.0] | 9.5 [8.5 to 10.0] | 9.0 [8.0 to 11.0]

31. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Sacrum, at Baseline
Description: Skin roughness was measured using the Visioscan VC98 (Courage+Khazaka, Cologne, Germany). It consists of a UV light camera and measures the skin surface profiles. Rmax (Maximum roughness) is the biggest roughness of the different segment roughness values.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 51.0 [42.5 to 56.0] | 47.5 [42.8 to 57.0] | 46.5 [38.5 to 53.5]

32. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Sacrum, After Two Hours Loading
Description: as for outcome 31
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 51.0 [45.5 to 59.0] | 50.0 [46.0 to 57.5] | 52.0 [43.5 to 58.5]

33. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Sacrum, 20 Min Off-loading
Description: as for outcome 31
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 57.0 [49.5 to 63.5] | 52.5 [45.5 to 65.0] | 52.0 [47.5 to 61.0]

34. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Heel, at Baseline
Description: as for outcome 25
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 48.5 [32.0 to 68.0] | 48.3 [36.1 to 59.4] | 51.5 [34.5 to 72.0]

35. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Heels, After Two Hours Loading
Description: as for outcome 25
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 50.5 [43.5 to 63.5] | 51.5 [45.0 to 72.0] | 51.0 [39.5 to 70.5]

36. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Heels, 20min Off-loading
Description: as for outcome 25
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 52.5 [46.0 to 73.0] | 59.5 [53.0 to 88.0] | 55.0 [40.0 to 58.5]

37. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Heels, at Baseline
Description: as for outcome 28
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 9.0 [7.5 to 13.5] | 9.8 [7.9 to 12.0] | 9.5 [7.0 to 15.5]

38. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Heels, After Two Hours Loading
Description: as for outcome 28
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 10.0 [7.5 to 12.0] | 10.0 [9.0 to 12.0] | 8.5 [7.5 to 13.0]

39. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Heels, 20 Min After Off-loading
Description: as for outcome 28
Time Frame: 20 min after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 10.5 [8.5 to 14.0] | 11.5 [9.5 to 17.0] | 9.0 [8.0 to 11.5]

40. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Heel, After Two Hours Loading
Description: as for outcome 31
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 67.5 [59.0 to 83.0] | 73.5 [57.0 to 100.5] | 67.5 [52.0 to 93.0]

41. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Heel, at Baseline
Description: as for outcome 31
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 63.5 [44.0 to 93.0] | 63.8 [46.6 to 79.5] | 70.0 [44.5 to 91.0]

42. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Heel, 20 Min After Off-loading
Description: as for outcome 31
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 71.5 [61.5 to 94.5] | 81.5 [69.0 to 110.5] | 70.0 [54.0 to 81.5]

43. Secondary Outcome: Skin Extensibility (Uf) in mm at the Sacrum, at Baseline
Description: Skin extensibility was measured using the Cutometer® MPA 580 and the corresponding software (Courage & Khazaka Electronic GmbH, Cologne, Germany).The measurements were conducted with a pressure of -450 mBar and a probe opening of 2 mm diameter and expressed in terms of total extensibility of the skin in mm (Uf, mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.32 [0.31 to 0.35] | 0.29 [0.26 to 0.33] | 0.32 [0.28 to 0.34]

44. Secondary Outcome: Skin Extensibility (Uf) in mm at the Sacrum, After Two Hours Loading
Description: Skin extensibility was measured using the Cutometer® MPA 580 and the corresponding software (Courage & Khazaka Electronic GmbH, Cologne, Germany).The measurements were conducted whit a pressure of -450 mBar and a probe opening of 2 mm diameter and expressed in terms of total extensibility of the skin in mm(Uf, mm).
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.34 [0.32 to 0.40] | 0.32 [0.28 to 0.37] | 0.35 [0.32 to 0.37]

45. Secondary Outcome: Skin Extensibility (Uf) in mm at the Sacrum, 20 Minutes After Off-loading
Description: Skin extensibility was measured using the Cutometer® MPA 580 and the corresponding software (Courage & Khazaka Electronic GmbH, Cologne, Germany).The measurements were conducted whit a pressure of -450 mBar and a probe opening of 2 mm diameter and expressed in terms of total extensibility of the Skin in mm (Uf, mm).
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.33 [0.30 to 0.38] | 0.31 [0.27 to 0.35] | 0.32 [0.30 to 0.37]

46. Secondary Outcome: Skin Extensibility (Uf) in mm at the Heel, at Baseline
Description: as for outcome 45
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.08 [0.07 to 0.12] | 0.08 [0.06 to 0.10] | 0.09 [0.08 to 0.10]

47. Secondary Outcome: Skin Extensibility (Uf) in mm at the Heel, After Two Hours Loading
Description: as for outcome 45
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.10 [0.08 to 0.12] | 0.10 [0.10 to 0.12] | 0.10 [0.08 to 0.12]

48. Secondary Outcome: Skin Extensibility (Uf) in mm at the Heel, 20 Minutes After Off-loading
Description: as for outcome 45
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.08 [0.07 to 0.12] | 0.09 [0.06 to 0.11] | 0.10 [0.08 to 0.12]

49. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Sacrum, at Baseline
Description: The elastic recovery (elastic recovery (Ur) / maximum extension (Uf)) of the skin was measured using the Cutometer® MPA 580 and the corresponding software (Courage & Khazaka Electronic GmbH, Cologne, Germany).The measurements were conducted whit a pressure of -450 mBar and a probe opening of 2 mm Diameter.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.55 [0.42 to 0.64] | 0.52 [0.46 to 0.64] | 0.57 [0.43 to 0.66]

50. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Sacrum, After Two Hours Loading
Description: as for outcome 49
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.55 [0.42 to 0.65] | 0.50 [0.42 to 0.66] | 0.44 [0.42 to 0.64]

51. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Sacrum, 20 Minutes After Off-loading
Description: as for outcome 49
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.52 [0.41 to 0.68] | 0.45 [0.37 to 0.66] | 0.51 [0.44 to 0.64]

52. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Heel, at Baseline
Description: as for outcome 49
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.36 [0.32 to 0.42] | 0.35 [0.33 to 0.39] | 0.35 [0.33 to 0.43]

53. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Heel, After Two Hours Loading
Description: as for outcome 49
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.35 [0.30 to 0.37] | 0.36 [0.32 to 0.40] | 0.38 [0.32 to 0.42]

54. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Heel, 20 Minutes After Off-loading
Description: as for outcome 49
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.34 [0.32 to 0.38] | 0.36 [0.33 to 0.38] | 0.35 [0.32 to 0.37]

55. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Sacrum, at Baseline
Description: The elastic function (Ur/Ue) of the skin was measured using the Cutometer® MPA 580 and the corresponding software (Courage & Khazaka Electronic GmbH, Cologne, Germany).The measurements were conducted whit a pressure of -450 mBar and a probe opening of 2 mm Diameter.
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.79 [0.54 to 0.90] | 0.78 [0.65 to 0.96] | 0.80 [0.67 to 0.97]

56. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Sacrum, After Two Hours Loading
Description: as for outcome 55
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.81 [0.65 to 0.87] | 0.70 [0.63 to 0.93] | 0.65 [0.56 to 0.90]

57. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Sacrum, 20 Minutes After Off-loading
Description: as for outcome 55
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.75 [0.56 to 0.92] | 0.66 [0.57 to 0.97] | 0.72 [0.59 to 0.80]

58. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Heel, at Baseline
Description: as for outcome 55
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.67 [0.64 to 0.77] | 0.68 [0.63 to 0.98] | 0.68 [0.62 to 0.85]

59. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Heel, After Two Hours Loading
Description: as for outcome 55
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.66 [0.58 to 0.79] | 0.70 [0.62 to 0.83] | 0.70 [0.62 to 0.81]

60. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Heel, 20 Minutes After Off-loading
Description: as for outcome 55
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.67 [0.61 to 0.79] | 0.67 [0.64 to 0.74] | 0.67 [0.61 to 0.75]

61. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Sacrum, at Baseline
Description: Epidermal moisture (measurement depth 0,5mm) was measured using MoistureMeterEpiD (Delfin Technologies Ltd.). The values are expressed in percentage of local tissue water (0 to 100 %).
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 41.0 [39.6 to 43.6] | 40.0 [36.5 to 42.0] | 41.0 [39.0 to 47.0]

62. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Sacrum, After Two Hours Loading
Description: as for outcome 61
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 44.5 [42.5 to 48.5] | 41.5 [40.5 to 47.5] | 43.5 [41.0 to 49.5]

63. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Sacrum, 20 Minutes After Off-loading
Description: as for outcome 61
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 44.5 [43.0 to 46.0] | 42.5 [39.5 to 46.5] | 44.0 [41.0 to 48.0]

64. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Heel, at Baseline
Description: as for outcome 61
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 25.5 [21.5 to 29.0] | 25.5 [21.5 to 30.0] | 24.0 [21.5 to 27.5]

65. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Heel, After Two Hours Loading
Description: as for outcome 61
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 28.0 [25.0 to 32.0] | 25.5 [25.0 to 27.5] | 28.0 [27.0 to 31.5]

66. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Heel, 20 Minutes After Off-loading
Description: as for outcome 61
Time Frame: 20 minutes after off-loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 25.5 [22.5 to 30.0] | 25.5 [23.5 to 28.0] | 25.5 [23.5 to 28.5]

67. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Sacrum
Description: Skin thickness was measured in μm (Metric) by Image Processing using Optical Coherence Tomography, OCT (Thorlabs, Lübeck, Germany).
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Groups:
- Standard Mattress: Basic foam: Standard mattress, Stryker, USA
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.09 [0.08 to 0.12]

68. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Sacrum
Description: as for outcome 67
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.08 [0.06 to 0.10]

69. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Heel
Description: as for outcome 67
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.43 [0.32 to 0.55]

70. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Heel
Description: as for outcome 67
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.45 [0.38 to 0.51]

71. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Sternum (Control- Area)
Description: as for outcome 67
Time Frame: baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.08 [0.06 to 0.09]

72. Secondary Outcome: Epidermal Thickness in μm (Metric) by Image Processing and Measurement at the Sternum (Control- Area)
Description: as for outcome 67
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Standard Mattress
Number analyzed (Participants) | 15
µm | 0.08 [0.07 to 0.09]

73. Secondary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Sternum (Control- Area), at Baseline
Description: TEWL was measured on sternum (control- area) using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany)
Time Frame: at baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 10.4 [9.3 to 11.8] | 9.8 [8.6 to 10.8] | 9.8 [8.7 to 12.3]

74. Secondary Outcome: Transepidermal Water Loss (TEWL) in g/m2/h on Sternum (Control- Area), After Two Hours Loading
Description: TEWL was measured on sternum (control- area) using the Tewameter TM300 (Courage & Khazaka, Cologne, Germany).
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: g/m2/h
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
g/m2/h | 8.3 [7.1 to 8.9] | 8.0 [7.2 to 8.7] | 8.1 [7.7 to 10.8]

75. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Sternum (Control- Area), at Baseline
Description: as for outcome 7
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 30.8 [29.9 to 31.2] | 30.7 [30.1 to 31.1] | 30.9 [30.4 to 31.2]

76. Secondary Outcome: Skin Surface Temperature in °C Per Skin Area at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 7
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: °C
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
°C | 29.9 [29.1 to 31.1] | 30.2 [29.7 to 30.9] | 30.6 [30.0 to 31.3]

77. Secondary Outcome: Erythema Index in Arbitrary Units at the Sternum (Control- Area), at Baseline
Description: as for outcome 13
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 317.7 [275.7 to 446.3] | 342 [266.9 to 417.9] | 390.2 [307.8 to 445.2]

78. Secondary Outcome: Erythema Index in Arbitrary Units at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 13
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 344.2 [305.0 to 425.9] | 350.2 [286.5 to 411.9] | 325.9 [280.5 to 482.5]

79. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Sternum (Control- Area), at Baseline
Description: as for outcome 19
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 48.1 [38.9 to 53.6] | 50.0 [41.4 to 60.9] | 47.0 [38.7 to 57.7]

80. Secondary Outcome: Stratum Corneum Hydration (SCH) in Arbitrary Units at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 19
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: arbitrary units
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
arbitrary units | 46.7 [34.1 to 50.5] | 43.7 [35.5 to 53.9] | 44.3 [31.7 to 62.8]

81. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Sternum (Control- Area), at Baseline
Description: as for outcome 61
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 50.0 [49.0 to 52.5] | 52.0 [44.5 to 55.5] | 51.5 [37.5 to 57.5]

82. Secondary Outcome: Epidermal Moisture Measurements Per Skin Area in Percentage (%) at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 61
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of tissue water content
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of tissue water content | 45.5 [41.0 to 55.0] | 51.5 [43.0 to 55.5] | 51.5 [47.5 to 56.0]

83. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Sternum (Control- Area), at Baseline
Description: as for outcome 25
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 36.5 [32.0 to 40.0] | 37.8 [31.5 to 42.9] | 35.0 [31.0 to 40.0]

84. Secondary Outcome: Skin Surface Mean Roughness (Rz) in μm at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 25
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 29.0 [26.0 to 32.5] | 28.5 [26.0 to 34.0] | 28.0 [23.5 to 32.0]

85. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Sternum (Control- Area), at Baseline
Description: as for outcome 28
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 8.0 [7.0 to 9.0] | 7.3 [7.0 to 8.5] | 8.5 [7.0 to 9.0]

86. Secondary Outcome: Skin Surface Mean Roughness (Ra) in μm at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 28
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 7.0 [6.0 to 9.0] | 7.0 [6.0 to 7.5] | 7.0 [6.0 to 8.0]

87. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Sternum (Control- Area), at Baseline
Description: as for outcome 31
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 48.5 [41.5 to 51.5] | 49.0 [41.5 to 56.6] | 44.5 [38.5 to 52.0]

88. Secondary Outcome: Skin Surface Maximum Roughness (Rmax) in µm at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 31
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: µm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
µm | 38.5 [34.0 to 42.0] | 38.5 [34.5 to 42.5] | 36.0 [30.5 to 41.5]

89. Secondary Outcome: Skin Extensibility (Uf) in mm at the Sternum (Control- Area), at Baseline
Description: as for outcome 45
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.34 [0.25 to 0.39] | 0.32 [0.28 to 0.37] | 0.36 [0.28 to 0.42]

90. Secondary Outcome: Skin Extensibility (Uf) in mm at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 45
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
mm | 0.32 [0.27 to 0.39] | 0.32 [0.24 to 0.34] | 0.37 [0.27 to 0.40]

91. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Sternum (Control- Area), at Baseline
Description: as for outcome 55
Time Frame: Baseline
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.59 [0.47 to 0.98] | 0.32 [0.28 to 0.37] | 0.70 [0.57 to 0.80]

92. Secondary Outcome: Skin Elastic Function (Ur/Ue) at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 55
Time Frame: after two hours loading
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: percentage of net elasticity
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
percentage of net elasticity | 0.71 [0.49 to 1.00] | 0.32 [0.24 to 0.34] | 0.68 [0.49 to 0.95]

93. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Sternum (Control- Area), at Baseline
Description: as for outcome 49
Time Frame: Baseline
Population: Cross-over trial with 15 female participants between 60 and 80 years, each of them lay on every of the three types of mattress.
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.42 [0.32 to 0.64] | 0.43 [0.31 to 0.57] | 0.47 [0.42 to 0.59]

94. Secondary Outcome: Elastic Recovery (Ur/Uf) at the Sternum (Control- Area), After Two Hours Loading
Description: as for outcome 49
Time Frame: after two hours loading
Population: as for outcome 93
Measure: Median (Inter-Quartile Range); unit: proportion of the elastic recovery
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
Number analyzed (Participants) | 15 | 15 | 15
proportion of the elastic recovery | 0.47 [0.33 to 0.66] | 0.48 [0.41 to 0.58] | 0.43 [0.38 to 0.61]

ADVERSE EVENTS:
Time Frame: Adverse event immediately or after loading of 2 hours on every of the three types of mattresses during each visit (three visits per subject, observation lasted up to 1 hour after each intervention) between September 2016 and March 2017 should be documented.
Arm/Group | Alternating Low Pressure Mattress | Reactive Support Surface | Standard Mattress
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT02930590/Prot_SAP_000.pdf